CLINICAL TRIAL: NCT03338660
Title: The Impact of Various Storage Techniques on Platelet Function
Brief Title: Platelet Function With Various Storage Techniques
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to begin study due to funding. PI has left organization.
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-XXXX-SIUHN
Record Dates: First submitted 2017-02-01; First posted 2017-11-09 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Platelet Dysfunction Due to Drugs
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: crossover study of various storage infusions techniques with each subject receiving various fluids aliquots.
Who Masked: Investigator, Outcomes Assessor
Masking Description: the assesor of platelet function and the PI will be blinded to group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (Placebo) (Placebo Comparator): Subjects will receive infusion of placebo (saline).
  Interventions: Biological: Placebo
- Platelet storage routine (Active Comparator): Subjects will receive infusion of platelets stored by routine method.
  Interventions: Biological: Infusion of Platelets
- Platelet storage experimental (Experimental): Subjects will receive infusion of platelets stored by a novel methodology.
  Interventions: Biological: Infusion of Platelets

INTERVENTIONS:
Biological: Infusion of Platelets — Platelets will be stored using novel, FDA approved, technique. Subjects will receive infusion of platelets stored by novel technique, routine storage, and placebo (saline).
  Other Names: Novel Storage Methodology
  Arms: Platelet storage experimental
Biological: Infusion of Platelets — Platelets will be stored using the routine platelet storage method. Subjects will receive infusion of platelets stored by routine storage method.
  Other Names: Routine Storage Method
  Arms: Platelet storage routine
Biological: Placebo — Subjects will receive infusion placebo (saline).
  Other Names: Placebo (Saline)
  Arms: Control (Placebo)

SUMMARY:
Platelet function will be tested in individuals on antiplatelet medications to determine the optimal storage methodology.

DETAILED DESCRIPTION:
Subjects will undergo administration of antiplatelet drugs and then will receive platelets stored in a variety of methods. Platelet function will be measured serially.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects

Exclusion Criteria:

* Pre existing antiplatelet drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-15 (Estimated); Primary Completion 2019-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in platelet function | 1 hour post-transfusion
  Frozen platelets will result in improvement in platelet function after transfusion.

IPD SHARING:
Plan to Share IPD: No